CLINICAL TRIAL: NCT05841238
Title: A Multiple Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Tablet and Capsule Formulations of LY3502970 in Healthy Overweight and Obese Participants
Brief Title: A Multiple Dose Study of LY3502970 in Healthy Overweight and Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18527; J2A-MC-GZGN (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Obese
MeSH Terms: conditions — Obesity | interventions — orforglipron

STUDY DESIGN:
Masking Description: Part A open label. Part B double blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3502970 (Part A) (Experimental): The multiple doses of LY3502970 administered orally either in tablet or capsule formulations.
  Interventions: Drug: LY3502970
- LY3502970 (Part B) (Experimental): The multiple doses of LY3502970 administered orally in tablet formulation.
  Interventions: Drug: LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally.

SUMMARY:
The main purpose of this study is to evaluate how much LY3502970 gets into the bloodstream and how long it takes the body to eliminate when administered orally as tablet and capsule formulations along with effect of food on LY3502970 in healthy overweight and obese participants. The study will also evaluate the safety and tolerability of LY3502970 in these participants. The study is conducted in two parts (part A and B) and will last up to 135 days including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are overtly healthy as determined by medical evaluation
* Participants with body mass index (BMI) of 27.0 kilograms per meter squared (kg/m²) or more
* Participants with a stable body weight, with 5% or less body weight gain or loss

Exclusion Criteria:

* Have any type of diabetes with hemoglobin A1c (HbA1c) level of 6.5% or greater or a fasting blood sugar over 120 milligram per deciliter (mg/dL)
* Obesity induced by other endocrine disorders, such as Cushing's syndrome or Prader-Willi syndrome
* Have known clinically significant gastric emptying abnormality
* Have undergone bariatric surgery (for example: Lap-Band, Gastric Bypass)
* Known self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or any form of thyroid cancer
* Have significant previous or current history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drug
* Have significant history of or currently have Major Depressive Disorder or psychiatric disorder within the last 2 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to the 24 Hour Time Point (AUC[0-24]) of LY3502970 | Predose up to 92 days postdose
  PK: AUC[0-24] of LY3502970
PK: Maximum Observed Concentration (Cmax) of LY3502970 | Predose up to 92 days postdose
  PK: Cmax of LY3502970
PK: Time to Maximum Observed Concentration (Tmax) of LY3502970 | Predose up to 92 days postdose
  PK: Tmax of LY3502970

SECONDARY OUTCOMES:
PK: AUC[0-24] of LY3502970 in fed state | Predose up to 92 days postdose
  PK: AUC[0-24] of LY3502970 in fed state
PK: Cmax of LY3502970 in fed state | Predose up to 92 days postdose
  PK: Cmax of LY3502970 in fed state
PK: Tmax of LY3502970 in fed state | Predose up to 92 days postdose
  PK: Tmax of LY3502970 in fed state

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - Labcorp Clinical Research LP, Dallas, Texas
  - LabCorp CRU, Inc., Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No